CLINICAL TRIAL: NCT02813850
Title: Impact of Home-based Oxygen Therapy on Maternal and Fetal Complications, in Pregnant Women With Sickle Cell Disease. A Randomized Multi-center Trial.
Brief Title: Oxygen Therapy and Pregnancy in Sickle Cell Disease
Acronym: DRO2G
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P140030; 2015-A01276-43 (Registry Identifier: ID RCB)
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; oxygen therapy; pregnancy; pregnancy in sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): standard medical care
- oxygen therapy (Experimental)
  Interventions: Device: oxygen therapy

INTERVENTIONS:
Device: oxygen therapy — Oxygen therapy early in the night (2L/min) during 4hours per days
  Arms: oxygen therapy

SUMMARY:
The purpose of this study is to assess the efficiency of the preventive oxygen therapy on the occurrence of vaso-occlusive complications, which last more than 24 hours and require hospitalisation, in women with sickle cell disease.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) corresponds to a group of inherited disorders with clinical manifestations resulting from the biochemical consequences of a single-base substitution of valine by glutamic acid at position 6 of the ß-hemoglobin (Hb) subunit (HbA [ß6val] to HbS [ß6glu]). When the oxygen tension is low, the solubility of HbS falls and the molecules polymerize. In turn, the intracellular formation of HbS polymers results in red blood cell (RBC) sickling. The aggregation of sickle cells is responsible for the vaso-occlusive crises (VOCs) that characterize SCD.

Thanks to improvements in the management of SCD patients, over 95% of affected infants survive to adulthood. Pregnancy is a high-risk situation for women with sickle cell disease, especially in the third trimester, during delivery and in the post-partum period. Conversely sickle cell disease can lead to pregnancy complications for both mother and fetus since maternal-fetal mortality remains elevated.

RBC transfusions and careful prevention of infections represent the only available treatments in this situation.

The complexity of this setting and the associated therapeutic strategy is further accentuated by the high frequency of post-transfusion side effects during SCD pregnancies, can indirectly affect the newborn by inducing hypoxia, and may ultimately prevent the woman from receiving further transfusions (RCOG, 2015) (Tuck et al, 1983). Post-transfusion complications constitute negative prognostic factors that affect both the mother's health and fetal development and thus increase the risk of premature death.

Another factor complicating the outcome of the pregnancy is the increase in oxygen demand in order to satisfy the increased metabolic requirements of the placenta and fetus. As the maternal oxygen reserve can be compromised during pregnancy for several reasons (such as the increased oxygen consumption, the SCD related anemia accentuated by the plasmatic increase), patients are particularly susceptible to hypoxemia - leading to the exacerbation of sickling events and SCD-related complications. (Hill & Pickinpaugh, 2008)(Thame et al, 2007)(Rathod et al, 2007a)(Cines et al, 1998)(Hassell, 2005)(Pantanowitz et al, 2000)(Rathod et al, 2007b) Moving from this observation, the first innovative approach introduced was the widespread use of prophylactic oxygen treatment at home. The rationale behind this change came from experiments on a murine model of SCD mice, in which a high-oxygen environment during pregnancy was associated with a lower prenatal fetal/maternal mortality rate (Ye et al, 2008). The absence of severe complications was also noticed in some women who could not be transfused (because of severe alloimmunization) and who were already receiving oxygen therapy at home before pregnancy.

Then a preliminary retrospective study was performed to evaluate the clinical benefit of the widespread use of prophylactic oxygen treatment at home. It indicates that this innovative treatment is safe and seems to be associated with a significant decrease in the transfusion rate in SCD patients during pregnancy.

These findings are encouraging, but they are preliminary and bias have to be taken into account. These results have to be confirmed by a randomized trial.

The project aim is to assess preventive oxygen therapy impact on women with sickle cell disease, their fetal and their newborn. Firstly, investigators want to assess preventive home-based oxygen therapy efficacy for preventing vaso-occlusive complications which last 24 hours and require a hospitalization. Secondly, they want to assess oxygen therapy impact on prevention and characteristics of obstetrical complications, prevention of neonatal complications, fetal and newborn's characteristics, type of medical care, transfusion balance sheet, way of transfusion and maternal, fetal and newborn tolerability of home-based oxygen therapy during pregnancy.

For this they propose to analyze 200 pregnant SCD women. 100 women in the first arm with standard medical care. 100 women in the second arm who will have home-based oxygen therapy early at night.

This study will be performed in 9 French hospitals. Blood samples of SCD women and blood cord will be drawn to monitor red cell adherence protein expression and function and their mechanic and adhesive properties.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women from 18 to 50 years old
* Maximal term: 20SA
* Patient with sickle cell disease
* Consent form signed by the patient
* Affiliated or beneficiary of a health insurance regimen and State Medical Aid.

Exclusion Criteria:

* Patients with transfusion restrictions
* Patients whose house can not receive the device
* Patients who have a weekly use of prophylactic oxygen therapy at home
* Patients who don't understand the operating instructions *Include patients with a doctor's prescription only. The portable oxygen concentrator will be removed from patients' home at the initiation visit prior to the overnight home oximetry test.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of at least one vaso-occlusive complication which last more than 24h | 30 days postpartum
  Painful vaso-occlusive episodes in bones, acute chest syndrome, ischemic stroke, cardiomyopathy, pulmonary hypertension, splenic and hepatic sequestration, death of the mother

SECONDARY OUTCOMES:
Occurrence of at least one vaso-occlusive complication which last more than 24h | 30 days postpartum
  Painful vaso-occlusive episodes in bones, acute chest syndrome, ischemic stroke, cardiomyopathy, pulmonary hypertension, splenic and hepatic sequestration, death of the mother
Occurrence of pregnancy-induced hypertension, pre-eclampsia, eclampsia | 20 months
Occurence of hospitalisation because of premature delivery risk | 20 months
Occurence of late miscarriage | 20 months
Occurence of Preterm (<35SA) and very preterm ( from 26 to 32SA) | 20 months
Type of delivery (vaginal, active, caesarean) | 20 months
Number of days hospitalisation postpartum | 20 months
Occurence of Neonatal complications ( respiratory distress, analgesics withdrawal symptom) | 20 months
Number of days of hospitalisation for the newborn | 20 months
Number of days of hospitalisation in resuscitation unit for the newborn | 20 months
Newborn weight | 20 months
Newborn size | 20 months
Newborn head circumference | 20 months
Apgar score assess 1 min after birth | 20 months
Apgar score assess 5 min after birth | 20 months
Apgar score assess 10 min after birth | 20 months
Perinatal and neonatal death | 20 months
pH of of the newborn | 20 months
Lactate of of the newborn | 20 months
Number of days using painkiller (level II and III) during pregnancy | 20 months
Number of urgent consultation | 20 months
Number of days of hospitalisation and hospitalisation in intensive care during pregnancy | 20 months
Stage of pregnancy at the first transfusion | 20 months
Total volume of transfusion during pregnancy | 20 months
Way of transfusion: simple, bleeding-transfusion, erythrocytapheresis | 20 months
Maternal, fetal and newborn tolerability of home-based oxygen therapy during pregnancy | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra BENACHI, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Laure JOSEPH, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Marina CAVAZZANA, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker Enfants-Malades (Public Hospitals of Paris), Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No